CLINICAL TRIAL: NCT04599062
Title: Neoadjuvant Intralesional Injection of Talimogene Laherparepvec With Concurrent Preoperative Radiation in Patients With Locally Advanced Soft Tissue Sarcomas
Brief Title: TVEC and Preop Radiation for Sarcoma (8 ml Dose)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Rieth (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, John Rieth, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504731 (8 milliliter dose)
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — talimogene laherparepvec; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Talimogene Laherparepvec in combination with radiotherapy-Phase I Cohort (Experimental): Talimogene Laherparepvec Dose Levels:
  Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Dose -1 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed every 2 weeks
  Interventions: Drug: Talimogene Laherparepvec; Radiation: Radiotherapy
- Talimogene Laherparepvec in combination with radiotherapy-Phase II Cohort (Active Comparator): Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Interventions: Drug: Talimogene Laherparepvec; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene Laherparepvec
Radiation: Radiotherapy — Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.

SUMMARY:
The purpose of this research study is to determine the safety and tolerability of talimogene laherparepvec when combined with radiation therapy.

Approximately 46 people will take part in this study conducted by investigators at the University of Iowa.

DETAILED DESCRIPTION:
This is a single-arm open-label phase Ib and phase II clinical study assessing the safety and relative efficacy of concurrent talimogene laherparepvec in combination with radiotherapy in patients with soft tissue sarcomas. Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery. Surgery will be performed 4-6 weeks from the end of radiation therapy to allow for resolution of acute toxicities per current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Histologically confirmed diagnosis of locally advanced STS that is unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate.

EXAMPLES:

* Resectable stage IIB, III, and IV disease that are not suitable for surgically resection alone due to inability to achieve clear margins.
* Including metastatic (stage IV) disease for which radiotherapy and surgical resection are indicated.
* Except certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma, bone sarcomas and myxoid liposarcomas (Grade 1).
* Previous treatment: prior systemic anti-cancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy are allowed provided therapy completed at least 1 year prior to enrollment.
* No prior Talimogene laherparepvec or tumor vaccines allowed.
* No prior radiation to the same tumor bed allowed.

  * Age ≥18 years.
  * Both men and women of all races and ethnic groups are eligible for this trial.
  * ECOG performance status ≤1.
  * Patient must have measurable disease:
* Tumor size at least ≥ 5 cm in the longest diameter as measured by CT scan or MRI for which radiation is feasible.

  * Patient must have injectable disease (direct injection or ultrasound guided).

Exclusion Criteria:

* Certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma bone sarcomas and low grade myxoid liposarcomas ( Grade 1).
* History or evidence of sarcoma associated with immunodeficiency states (e.g.: Hereditary immune deficiency, HIV, organ transplant or leukemia).
* Subjects with retroperitoneal and visceral sarcoma.
* History or evidence of gastrointestinal inflammatory bowel disease (ulcerative colitis or Crohn's disease) or other symptomatic autoimmune disease including, inflammatory bowel disease, or history of any poorly controlled or severe systemic autoimmune disease (i.e., rheumatoid arthritis, systemic lupus erythematosus, scleroderma, type I diabetes, or autoimmune vasculitis).
* History of other malignancy within the past 3 years except treated with curative intent and no known active disease present and has not received chemotherapy for ≥ 1 year before enrollment/randomization and low risk for recurrence.
* History of prior or current autoimmune disease.
* History of prior or current splenectomy or splenic irradiation.
* Active herpetic skin lesions
* Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use.
* Any non-oncology vaccine therapies used for the prevention of infectious disease within 28 days prior to enrollment and during treatment period.
* Concomitant treatment with therapeutic anticoagulants such as warfarin. Patients on therapeutic low molecular weight heparin may be allowed provided the dose can be safely held as per the treating investigator on the morning of scheduled intratumoral injection and can be resumed 12 hours after the procedure
* Known human immunodeficiency virus (HIV) disease (requires negative test for clinically suspected HIV infection).
* Acute or chronic hepatitis B or hepatitis C infection (requires negative test for clinically suspected hepatitis B or hepatitis C infection).
* Evidence of hepatitis B -

  1. Positive HBV surface antigen (indicative for chronic hepatitis B or recent acute hepatitis B).
  2. Negative HBV surface antigen but positive HBV total core antibody (indicative for resolved hepatitis B infection or occult hepatitis B) and detectable copies of HBV DNA by PCR (detectable HBV DNA copies suggest occult hepatitis B).
* Evidence of hepatitis C -

  1. Positive HCV antibody and positive HCV RNA by PCR (undetectable RNA copies suggest past and resolved hepatitis C infection).
* Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment.
* Female subjects of childbearing potential or male subjects who are unwilling to use 2 highly effective methods of contraception during study treatment and through 3 months after the last dose of study treatment. See Section 7.5 for more details.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
* Other investigational procedures while participating in this study that could affect the primary objective of the study as determined by the PI are excluded.
* Subject previously has entered this study.
* Patients who are receiving any other investigational agents.
* Evidence of CNS metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talimogene laherparepvec.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients on or requiring immunosuppressive therapies.
* Any of the following laboratory abnormalities:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count (ANC) < 1500 per mm3
  * Platelet count < 100,000 per mm3
  * Total bilirubin > 1.5 × ULN
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN
  * Alkaline phosphatase > 2.5 × ULN
  * PT (or INR) and PTT (or aPTT) > 1.5 × ULN
  * Creatinine > 2.0 × ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2028-02-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Rieth, MD, Principal Investigator — University of Iowa Holden Comprehensive Cancer Center
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Talimogene Laherparepvec in Combination With Radiotherapy-Phase I: Talimogene Laherparepvec Dose Levels:
  Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
- Talimogene Laherparepvec in Combination With Radiotherapy-Phase II: Talimogene Laherparepvec Dose Level:
  Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec in Combination With Radiotherapy-Phase I | Talimogene Laherparepvec in Combination With Radiotherapy-Phase II
Started | 6 | 2
Completed | 5 | 2
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Talimogene Laherparepvec in Combination With Radiotherapy-Phase I: Talimogene Laherparepvec in combination with radiotherapy Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Talimogene Laherparepvec: Talimogene Laherparepvec
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
- Total: Total of all reporting groups
Arm/Group | Talimogene Laherparepvec in Combination With Radiotherapy-Phase I | Talimogene Laherparepvec in Combination With Radiotherapy-Phase II | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 5 | 0 | 5
Age, Continuous [Mean (Full Range); unit: years] | 72 [63 to 81] | 44 [34 to 53] | 65 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as any of the following talimogene laherparepvec-related toxicity or related to the combination of talimogene laherparepvec and radiation therapy during treatment and up to 4 weeks after the last talimogene laherparepvec injection: Grade 3 or greater immune-mediated adverse events, Grade 3 or greater allergic reactions, any grade plasmacytoma, any other unexpected grade 3 or greater hematologic or non-hematologic toxicity, with the exceptions of: any grade of alopecia, expected radiation related skin toxicity of any grade, Grade 3 arthralgia or myalgia, brief (< 1 week) grade 3 fatigue, Grade 3 fever, Grade 3 diarrhea or vomiting responding to supportive case.
Time Frame: 14 weeks
Population: 6 participants enrolled in the Phase 1 portion (Talimogene Laherparepvec Dose 0) and completed treatment, radiation, and surgical resection.
Measure: Count of Participants; unit: Participants
Groups:
- Talimogene Laherparepvec in Combination With Radiotherapy-Phase I Cohort: Talimogene Laherparepvec in combination with radiotherapy
  Talimogene Laherparepvec Dose Levels:
  Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
Arm/Group | Talimogene Laherparepvec in Combination With Radiotherapy-Phase I Cohort
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Pathologic Tumor Necrosis Rate
Description: Pathologic tumor necrosis rate is defined as the percentage of subjects with pathologic tumor necrosis ≥ 90%.
Time Frame: 14 weeks
Population: 8 participants received Dose Level 0 and were included in the analysis for pathologic tumor necrosis
Measure: Count of Participants; unit: Participants
Groups:
- Talimogene Laherparepvec in Combination With Radiotherapy: Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Talimogene Laherparepvec: Talimogene Laherparepvec
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
Arm/Group | Talimogene Laherparepvec in Combination With Radiotherapy
Number analyzed (Participants) | 8
Participants | 4

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of patients with a confirmed complete or partial response per RECIST v1.1.
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: 2 Year Progression-Free Survival
Description: Progression-free survival is defined as the time from treatment initiation to the date of first documentation of disease progression or death due to any cause. Otherwise, patients are censored at the date of last radiographic assessment for progression.
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: 2 Year Overall Survival
Description: Overall survival is defined as the time from treatment initiation to death due to any cause. Patients still alive are censored at last date known to be alive.
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information regarding the occurrence of adverse events was collected from the time the subject signed the informed consent form and throughout their participation in the study, through a period of 30 days after the last dose of study drug, up to 14 weeks.
Groups:
- Talimogene Laherparepvec in Combination With Radiotherapy-Phase I: Talimogene Laherparepvec in combination with radiotherapy
  Talimogene Laherparepvec Dose Levels:
  Dose 0 = talimogene laherparepvec up to 8.0 mL of 108 PFU/mL dosed weekly
  Talimogene Laherparepvec: Talimogene Laherparepvec
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
Arm/Group | Talimogene Laherparepvec in Combination With Radiotherapy-Phase I | Talimogene Laherparepvec in Combination With Radiotherapy-Phase II
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talimogene Laherparepvec in Combination With Radiotherapy-Phase I (N=6) | Talimogene Laherparepvec in Combination With Radiotherapy-Phase II (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders and administration site conditions) | 5 (7) | 2 (2)
Edema limbs (General disorders and administration site conditions) | 1 (1) | 1 (1)
Fatigue (General disorders and administration site conditions) | 5 (6) | 0 (0)
Fever (General disorders and administration site conditions) | 3 (5) | 2 (4)
Flu like symptoms (General disorders and administration site conditions) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders and administration site conditions) | 0 (0) | 1 (1)
Pain (General disorders and administration site conditions) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 (5) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment halted prematurely due to funding. Participants are being followed for secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT04599062/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04599062/ICF_001.pdf